CLINICAL TRIAL: NCT03717779
Title: Contribution of Pulmonary Ultrasonography in the Diagnosis of Acute Heart Failure (AHF) in Patients Admitted to Emergency Department (ED) for Dyspnea
Brief Title: Contribution LUS in the Diagnosis of Acute Heart Failure (AHF) in Patients Admitted to the ED
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Pr. Semir Nouira, University of Monastir
Other Study IDs: Lung Ultra Sound (LUS)
Record Dates: First submitted 2018-07-06; First posted 2018-10-24 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Dyspnea; Cardiac
Keywords: Lung ultrasound,; heart failure; diagnosis; accuracy
MeSH Terms: conditions — Dyspnea; Heart Failure; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HF/HFpEF: patients with heart failure with a preserved ejection fraction(HFpEF) perform LUS
  Interventions: Diagnostic Test: lung ultrasound
- HF/HFrEF: patients with heart failure with a reduced ejection fraction(HFrEF) perform LUS
  Interventions: Diagnostic Test: lung ultrasound

INTERVENTIONS:
Diagnostic Test: lung ultrasound — we perform a lung ultrasound to all the patients admitted for dyspnea independantly from the final diagnosis

SUMMARY:
This study assesses the potential of lung ultrasonography to diagnose heart failure.

DETAILED DESCRIPTION:
Dyspnea is one of the most distressing situations for the patient . Emergency cases do not always present in conditions that are ideal for immediate diagnosis, which sometimes compromises outcome. Physical examination, laboratory findings and radiography are imperfect, resulting in a need for sophisticated test results that delay management.

Lung ultrasonography is becoming a standard tool in critical cases in the ED.

the investigators aim to perform ultrasonography on consecutive patients admitted to the ICU with dyspnea, comparing lung ultrasonography results on initial presentation with the final diagnosis by the ICU team.

Three items were assessed: artifacts (horizontal A lines or vertical B lines indicating interstitial syndrome), lung sliding, and alveolar consolidation and/or pleural effusion, these items were grouped to assess ultrasound profiles.

This study assesses the potential of lung ultrasonography to diagnose heart failure.

ELIGIBILITY:
Inclusion Criteria:

* non traumatic dyspnea with the final diagnosis of heart failure

Exclusion Criteria:

* coma,
* shock,Mechanical Ventilation,
* vasopressor drugs
* arrhythmia serious and sustained,
* non consent

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients admitted to the ED with acute dyspnea, with the final diagnosis of heart failure by the ICU team
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
the accuracy of LUS in the diagnosis of heart failure | 0 days
  the accuracy of LUS in the diagnosis of heart failure measured by sensitivity ,specificity, and area under the roc curve

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, PHD, Principal Investigator — University hospital of Monastir
Locations (1):
- Emergency department of university hospital Fattouma Bourguiba of Monastir, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Msolli MA, Sekma A, Marzouk MB, Chaabane W, Bel Haj Ali K, Boukadida L, Bzeouich N, Gannoun I, Trabelssi I, Laaouiti K, Grissa MH, Beltaief K, Dridi Z, Belguith A, Methamem M, Bouida W, Boukef R, Boubaker H, Nouira S; GREAT Network. Bedside lung ultrasonography by emergency department residents as an aid for identifying heart failure in patients with acute dyspnea after a 2-h training course. Ultrasound J. 2021 Feb 9;13(1):5. doi: 10.1186/s13089-021-00207-9. PMID 33559777
- See also: official department website — http://www.urgencemonastir.com